CLINICAL TRIAL: NCT03226743
Title: Collaborative and Stepped Care in Mental Health by Overcoming Treatment Sector Barriers: A Cluster-randomized Controlled Trial (COMET)
Brief Title: Collaborative and Stepped Care in Mental Health (COMET)
Acronym: COMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Center for Health Care Research Hamburg (Unknown); Hamburg Center for Health Economics (Other)
Responsible Party: Principal Investigator, Prof. Dr. Martin Härter, Prof. Dr. med Dr. phil. Dipl. Psych., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01GY1602
Record Dates: First submitted 2017-07-10; First posted 2017-07-24 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Depressive Disorder; Anxiety Disorder; Somatoform Disorder; Alcohol Use Disorder
Keywords: stepped and collaborative care; cluster-randomized controlled trial; health services research; evidence-based medicine; complex intervention; guideline implementation; collaborative network
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Somatoform Disorders; Alcoholism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): collaborative and stepped care model for depressive, anxiety, somatoform and/or alcohol abuse disorders within a multiprofessional network
  Interventions: Other: collaborative and stepped care model
- Control Group (No Intervention): treatment as usual in German health care system

INTERVENTIONS:
Other: collaborative and stepped care model — Including elements:
  * collaborative and stepped care of patients with mental disorders
  * treatment in a multiprofessional network consisting of primary care physicians, psychologists, psychiatrists and inpatient facilities
  * initial training of participating health care providers
  * formalized and standardized screening procedure for early recognition of depressive, anxiety, somatoform and alcohol abuse disorders
  * formalized ICD-diagnostics
  * guideline-oriented treatment recommendations
  * bibliotherapy or internet-based self-help for patient with mild to moderate disorders
  * online referral platform
  * case management for patients with severe disorders
  * systematic and regular monitoring
  * regular quality circles for participating health care providers
  Arms: Intervention Group

SUMMARY:
The aims of COMET are the implementation and evaluation of effectiveness and cost-effectiveness as well as processes of a collaborative and stepped care model for depressive, anxiety, somatoform and/or alcohol abuse disorders within a multiprofessional network in comparison to routine care. In a cluster-randomized controlled effectiveness trial 570 patients will be recruited by 38 general practitioner practices and followed with a prospective survey at four time points. The primary outcome is the change in health-related quality of life from baseline to 6-months follow-up. Secondary outcomes include disorder-specific symptom burden, response, remission, functional quality of life, cost-effectiveness, evaluation of processes and other clinical and psychosocial variables.

DETAILED DESCRIPTION:
Aims are a) the implementation and outcome evaluation, b) the process evaluation, and c) the analysis of the cost-effectiveness of an innovative collaborative and stepped care model for patients with depressive, anxiety, somatoform and/or alcohol abuse disorders.

Its novelty is the integration of these four disorders into one model. This approach is based on a) the high comorbidity between these disorders, b) the fact that they share a common etiological and diag-nostic basis, c) that similar evidence-based treatment options exist for them (e.g., self-help and psychoeducation, psychotherapy, pharmacotherapy), and d) that health care providers need to manage them together very often.

The conceptual basis follows the principles of evidence-based medicine with a specific focus on guideline implementation and the principles of patient-centered care including access, coordination and continuity of care, patient information, patient involvement and empowerment. Based on a multi-professional cooperation of health care providers across different care sectors an integrated health care network consisting of general practitioners (GPs), mental health specialists (psychiatrists, psychotherapists) and inpatient facilities will be established. Evidence-based clinical practice guidelines and pathways of care with treatment options of varying intensity form the clinical and procedural basis of the network, including low-intensity treatments and e-mental health technologies.

The study is planned as a randomized controlled effectiveness trial of a consecutive sample of patients with depressive and/or anxiety and/or somatoform and/or alcohol abuse disorders drawn from primary care (GP practices) and followed with a prospective survey at four time points. The study is intended to recruit a total of 570 patients from 38 GP practices. A cluster-randomization at the level of participating GP practices divides GPs into the intervention group, where patients are treated within a multi-professional collaborative and stepped care approach (including low-intensity treatments, direct access to mental health specialists, inpatient care etc., COMET), and the control group, where patients receive standard care (treatment as usual, TAU). Data collection is carried out with questionnaires as well as telephone interviews at four time-standardized measurement points within one year (baseline, 3, 6, 12 and 24 months). Additionally, independent research assistants perform standardized diagnostic interviews (CIDI) with patients at baseline to allow an assessment of diagnostic validity.

The main research hypothesis is that the COMET model is more effective than TAU. Primary outcome is the change in health-related quality of life measured by the SF-36 mental health score from baseline to 6-months follow-up. Secondary outcomes include symptom burden of depressive, generalized anxiety, panic, somatoform and alcohol abuse syndromes (PHQ-9; GAD-7; PHQ-15; PHQ panic and alcohol abuse syndrome module; SSD-12), disorder-specific response and remission, functional quality of life (EQ-5D-5L), duration of untreated illness, and other clinical and psychosocial variables (outcome evaluation, Work Package 1). Furthermore, direct and indirect costs and the incremental cost-effectiveness ratio will be assessed (economic evaluation, Work Package 2). Finally, feasibility and acceptance of the COMET model as well as of the different treatment components are assessed, including the implementation process (process evaluation, Work Package 3). To this end, semi-structured interviews will be conducted at two measurement points, supplemented by standardized surveys among involved patients and providers.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are a minimum age of 18, informed consent and one or more of the following positive ICD-10-diagnoses: depressive episode (F32), recurrent depressive disorder (F33), dysthymia (F34.1), agoraphobia (F40.0), social phobia (F40.1), panic disorder (F41.0), generalized anxiety disorder (F41.1), mixed anxiety and depressive disorder (F41.2), somatoform disorders (F45), and/or mental and behavioral disorders due to use of alcohol (F10.1, F.10.2)

Exclusion Criteria:

* Patients with insufficient knowledge of the German language, an acute psychosis or a health situation that does not allow questionnaire completion or patients already receiving current in- or outpatient psychiatric or psychotherapeutic care are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
change in health-related quality of life | from baseline to 6 months and 12 and 24 months after baseline
  measured with the Short Form Health Survey SF-36 mental health score

SECONDARY OUTCOMES:
change in disorder-specific symptoms: depression | from baseline to 6 months and 12 and 24 months after baseline
  measured on the major depressive module of the Patient Health Questionnaire PHQ: PHQ-9
change in disorder-specific symptoms: panic | from baseline to 6 months and 12 and 24 months after baseline
  measured on the panic module of the Patient Health Questionnaire PHQ: PHQ-panic module
change in disorder-specific symptoms: generalized anxiety | from baseline to 6 months and 12 months and 24 months after baseline
  measured on the generalized anxiety module of the Patient Health Questionnaire PHQ: GAD-7
change in disorder-specific symptoms: somatoform syndrome PHQ | from baseline to 6 months and 12 and 24 months after baseline
  measured on the somatoform module of the Patient Health Questionnaire PHQ: PHQ-15
change in disorder-specific symptoms: somatoform syndrome SSD-12 | from baseline to 6 months and 12 and 24 months after baseline
  measured on the Somatic Symptom Disorder-B SSD-12
change in disorder-specific symptoms: alcohol abuse disorder | from baseline to 6 months and 12 and 24 months after baseline
  measured on the Alcohol Use Disorders Identification Test: AUDIT
cost effectiveness: direct costs | from baseline to 6 months and 12 and 24 months after baseline
  will be assessed based on health care utilization, reduced productivity at work and work loss days measured by a modified version the Client Sociodemographic and Service Receipt Inventory (CSSRI). For the monetary valuation of resources, unit costs will be applied.
cost effectiveness: indirect costs | from baseline to 6 months and 12 and 24 months after baseline
  will be assessed based on health care utilization, reduced productivity at work and work loss days measured by a modified version the Client Sociodemographic and Service Receipt Inventory (CSSRI). Indirect costs will be calculated based on the human capital approach.
cost effectiveness: health effects | from baseline to 6 months and 12 and 24 months after baseline
  quality-adjusted life years (QALYs) will be calculated based on utilities derived from the EQ-5D-5L questionnaire
cost effectiveness: incremental cost-effectiveness | from baseline to 6 months and 12 and 24 months after baseline
  incremental cost-effectiveness ratios (ICER) will be calculated
cost effectiveness: acceptability | from baseline to 6 months and 12 and 24 months after baseline
  Cost-effectiveness acceptability curves (CEAC) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Härter, Prof. Dr. Dr., Principal Investigator — Center for Psychosocial Medicine, Department of Medical Psychology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany
Locations (1):
- University Medical Center Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grochtdreis T, Heddaeus D, Seeralan T, Maehder K, Porzelt S, Daubmann A, Pepic A, Lowe B, Rosenkranz M, Schafer I, Scherer M, Schulte B, von dem Knesebeck O, Weigel A, Wegscheider K, Werner S, Zapf A, Zimmermann T, Dirmaier J, Harter M, Konig HH, Dams J. Cost-utility analysis of a collaborative and stepped care model in patients with mental disorders in German primary care (the COMET study). BMC Psychiatry. 2025 Oct 13;25(1):973. doi: 10.1186/s12888-025-07428-5. PMID 41083989
- [Derived] Maehder K, Werner S, Weigel A, Lowe B, Heddaeus D, Harter M, von dem Knesebeck O. How do care providers evaluate collaboration? - qualitative process evaluation of a cluster-randomized controlled trial of collaborative and stepped care for patients with mental disorders. BMC Psychiatry. 2021 Jun 8;21(1):296. doi: 10.1186/s12888-021-03274-3. PMID 34098913
- [Derived] Weigel A, Maehder K, Witt M, Lowe B. Psychotherapists' perspective on the treatment of patients with somatic symptom disorders. J Psychosom Res. 2020 Nov;138:110228. doi: 10.1016/j.jpsychores.2020.110228. Epub 2020 Aug 29. PMID 32896756
- [Derived] Maehder K, Lowe B, Harter M, Heddaeus D, von dem Knesebeck O, Weigel A. Psychotherapists' perspectives on collaboration and stepped care in outpatient psychotherapy-A qualitative study. PLoS One. 2020 Feb 5;15(2):e0228748. doi: 10.1371/journal.pone.0228748. eCollection 2020. PMID 32023303
- [Derived] Heddaeus D, Dirmaier J, Brettschneider C, Daubmann A, Grochtdreis T, von dem Knesebeck O, Konig HH, Lowe B, Maehder K, Porzelt S, Rosenkranz M, Schafer I, Scherer M, Schulte B, Wegscheider K, Weigel A, Werner S, Zimmermann T, Harter M. Study protocol for the COMET study: a cluster-randomised, prospective, parallel-group, superiority trial to compare the effectiveness of a collaborative and stepped care model versus treatment as usual in patients with mental disorders in primary care. BMJ Open. 2019 Nov 24;9(11):e032408. doi: 10.1136/bmjopen-2019-032408. PMID 31767595
- [Derived] Maehder K, Lowe B, Harter M, Heddaeus D, Scherer M, Weigel A. Management of comorbid mental and somatic disorders in stepped care approaches in primary care: a systematic review. Fam Pract. 2019 Jan 25;36(1):38-52. doi: 10.1093/fampra/cmy122. PMID 30535053